CLINICAL TRIAL: NCT00964405
Title: Phase I Study of GSK233705- A Randomised, Double Blind, Placebo-controlled, 2-parts Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Single and Repeat Inhaled Doses of GSK233705 From a Novel Dry Powder Device in Healthy Japanese Male Subjects -
Brief Title: Phase I Study of GSK233705 in Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 112016
Record Dates: First submitted 2009-08-13; First posted 2009-08-24 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- LAMA (Experimental): After randomization subject will inhale either GSK233705 50, 100 or 200 microgram once daily for 7 days.
  Interventions: Drug: GSK233705
- Placebo (Placebo Comparator): After randomization subjects will inhale placebo once daily for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK233705 — Inhaled Long acting muscarinic receptor antagonist
  Arms: LAMA
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This is a randomised, double blind, placebo-controlled, 2-parts study to investigate the safety, tolerability, and pharmacokinetics of single and repeat inhaled doses of GSK233705 from a novel dry powder device in healthy Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese healthy male subjects aged between 20 and 64 years of age inclusive. Healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history, physical examination, laboratory studies, and other tests.
2. Body weight ≥ 50kg and BMI within the range 18.50-25.00kg/m2 inclusive.
3. Non-smokers (never smoked or not smoking for >6 months with <10 pack years history (Pack years = (cigarettes per day smoked/20) x number of years smoked))
4. Normal spirometry (FEV1 ≥ 80% of predicted, FEV1/FVC ≥ 70%).
5. Clinical laboratory tests data obtained at screening meet the following:

   AST(GOT), ALT(GPT), total-bilirubin: below the upper limit of the normal ranges
6. Normal 12-lead EGC finding at screening; QTc interval <450msec
7. A mean blood pressure lower than 140/90mmHg at screening.
8. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
9. Capable of using the novel dry powder inhaler.

Exclusion Criteria:

1. The subject has any clinically relevant abnormality on medical examination, vital sign, clinical laboratory test or medical history at screening in the medical opinion of the investigator or the subject has a medical history that is not considered as eligible for inclusion in this study by the investigator.
2. The subject is currently participating in another clinical study or post-marketing study in which the subject is or will be exposed to an investigational or a non-investigational drug or device.
3. The subject has participated in a clinical study with an investigational or a non-investigational drug or device during the previous 4 months.
4. A history of breathing problems (i.e. history of asthmatic symptomatology, asthma in childhood).
5. The subject has a known allergy or hypersensitivity to ipratropium bromide, tiotropium, atropine and any of its derivatives.
6. The subject has a known allergy or hypersensitivity to milk protein or the excipients lactose monohydrate and magnesium stearate.
7. The subject has a history or current conditions of drug abuse or alcoholism.
8. History of regular alcohol consumption exceeding on average, 14 drinks/week (1 drink=5 ounces (150mL) of wine or 350mL of beer or 1.5 ounces (45mL) of 80 proof distilled spirits) within 6 month of screening.
9. The subject is positive for urine drug screening.
10. The subject is positive for syphilis, HBs antigen, HCV antibody, HIV antibody, HTLV-1 antibody.
11. The subject has donated a unit of blood ">400mL" within the previous 4 months or ">200mL" within the previous 1 month.

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-09-20 (Actual); Primary Completion 2008-12-20 (Actual); Study Completion 2008-12-20 (Actual)

PRIMARY OUTCOMES:
Safety：adverse events, vital sign, ECGs, and clinical laboratory test
PK：Cmax, tmax and AUC(0-t)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fukuoka, Japan

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Results for study 112016 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/112016?search=study&search_terms=112016#rs